CLINICAL TRIAL: NCT06956300
Title: Grit Against Cognitive Decline in Aging and Preclinical Alzheimer's Disease
Brief Title: TMS for Cognitive Decline in Aging and Preclinical AD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Alexandra Touroutoglou, Assistant Professor of Neurology, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2023A009489
Record Dates: First submitted 2025-04-14; First posted 2025-05-04 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-04

CONDITIONS: Prodromal Alzheimer's Disease; Preclinical Alzheimer's Disease; Healthy Aging; Cognitive Decline
Keywords: Transcranial Magnetic Stimulation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TMS (Experimental): All participants will receive the same study interventions in a within-subject crossover design.
  Interventions: Device: Active rTMS
- Sham TMS (Sham Comparator): All participants will receive the same study interventions in a within-subject crossover design.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Active rTMS — All study participants will receive one block of ACTIVE rTMS. Each block will consist of daily sessions of active rTMS delivered to the left dorsolateral prefrontal cortex over ten days (Monday through Friday).
  Arms: Active TMS
Device: Sham rTMS — All study participants will receive one block of SHAM rTMS. Each block will consist of daily sessions of SHAM rTMS delivered to the left dorsolateral prefrontal cortex over ten days (Monday through Friday).
  Arms: Sham TMS

SUMMARY:
In this research study we want to learn more about the effects of non-invasive brain stimulation on motivation, memory, and brain-network function in cognitively unimpaired older adults and individuals with preclinical Alzheimer's disease.

This study will use a form of non-invasive brain stimulation called repetitive Transcranial Magnetic Stimulation (rTMS). rTMS will slightly alter activity in an area of your brain that controls cognition. Changes resulting from this stimulation will be measured with behavioral tests, as well as by taking brain images with Magnetic Resonance Imaging (MRI).

Participants will come in for one baseline visit followed by 10 days of daily rTMS study visits (Monday through Friday) and an evaluation visit. Then, there will be a 2-week break. After this break, they will return for another baseline visit, an additional 10 days of rTMS, and a final evaluation visit.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 40-99
2. Native English speakers
3. Willing and able to consent to the protocol and undergo imaging and neuropsychological testing at the specified time points
4. Cognitively normal older adults and individuals with preclinical Alzheimer's disease will be included.

Exclusion Criteria:

1. History of head trauma involving loss of consciousness or alteration in consciousness
2. Another major neurologic or psychiatric condition
3. Known presence of a structural brain lesion (e.g. tumor, cortical infarct)
4. Any contraindication to MRI, such as presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments, or foreign objects in the eyes, skin, or body
5. Longstanding premorbid history (i.e. longer than 10 years) of alcohol or substance abuse with continuous abuse up to and including the time that the symptoms leading to clinical presentation developed
6. Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the study protocol.
7. Unwilling to return for follow-up, undergo neuropsychological testing, TMS, and MR imaging
8. History of unprovoked seizures (i.e., seizures that occur in the absence of a clear provocation such as hyponatremia, hypoglycemia, etc.).
9. Subjects who have a first degree relative (e.g., father, mother or sibling) with a seizure disorder.
10. Subjects currently taking, or plan to take, medications which are highly epileptogenic. These include: clozapine, high doses of bupropion (i.e., greater than 400mg daily), diphenhydramine, cyclosporine, isoniazid, imipenem, chloroquine, tramadol and theophylline.

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in motivation | Baseline and post-treatment Day 11
  This will be measured by ratings of grit on a 5-point scale using the Grit Scale (Duckworth, et al., 2007).
Changes in Brain Network Connectivity | Baseline and post-treatment Day 11
  This will include changes in resting-state functional connectivity measured with functional Magnetic Resonance Imaging (fMRI)
Changes in Memory | Baseline and Post-Treatment Day 11
  This will be measured with an associative memory task

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No